CLINICAL TRIAL: NCT01606410
Title: The Impact of Age and Fitness on Endothelial Reperfusion Injury and the Ability of Ischemic Preconditioning to Prevent This Injury
Brief Title: The Impact of Age and Fitness on Reperfusion Injury and Ischemic Preconditioning to Prevent This Injury
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRI-IPC-aging
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- young, sedentary
  Interventions: Other: IPC
- young, active
  Interventions: Other: IPC
- old, sedentary
  Interventions: Other: IPC
- old, active
  Interventions: Other: IPC

INTERVENTIONS:
Other: IPC — repeated cuff inflation (220 mmhg) around an upper limb for 5 minutes, followed by 5 minutes of reperfusion (repeated 4 times)

SUMMARY:
Rationale: Ischaemic preconditioning (IP) refers to the reduction of ischemia-reperfusion injury induced by a brief preceding period of ischemia. Also the arterial endothelium can be protected by IP. Several studies performed in animals and humans have demonstrated that the protective effects of IP are attenuated with aging. However, no previous study directly examined the underlying mechanisms of this observation. Possibly, the reduced protective effect of IP with aging relates to a direct effect on the endothelium, consequently leading to an attenuated ability of IP to prevent endothelial dysfunction after ischaemia reperfusion injury.

Several previous studies failed to demonstrate the ability of pharmacological stimuli to mimic the beneficial effects of IP in aged vessels. Restoration of the age-related reduction in effectiveness of IP may be possible through exercise training. In aged animals, physical training restores the efficacy of ischemic preconditioning. Indirect evidence indicates that physical activity, independent of other cardiovascular risk factors, protects against a occurrence as well as the severity of a myocardial infarction in humans. Although this suggests that physical activity may beneficially influence the age-related reduction in IP, no previous study provided direct evidence for this hypothesis.

Objective: To examine the impact of age and physical fitness on the ability of ischaemic preconditioning to protect endothelial damage in response to ischaemia reperfusion injury in healthy humans. A secondary objective is to explore the role of Toll-like receptor (TLR) signalling in the induction of IP in young and old subjects.

DETAILED DESCRIPTION:
Cardiovascular disease has become a worldwide burden. In the Netherlands over 40.000 persons die annually due to coronary artery disease, either acute myocardial infarction or heart failure.1 Through plaque formation and negative vascular remodelling, significant stenotic lesions develop in the coronary arteries that subsequently limit coronary blood flow and ultimately can cause ischemic events. Reperfusion therapy (either pharmacologic, endovascular or surgical) is mandatory for salvage of ischemic tissue. However, during reperfusion several deleterious events take place causing further damage. Murry found that ischemia and reperfusion injury (IR-injury) could be reduced by a phenomenon called ischemic preconditioning.2 Short lasting repetitive episodes of ischemia prior to an ischemic event can induce tissue tolerance against IR-injury.

After discovery of this phenomenon, ample research has been devoted to elucidation of the underling protective mechanism, but also factors that improve or impair the ability of this phenomenon to protect arteries against ischaemia reperfusion injury. Several studies performed in animals and humans have demonstrated that the protective effects of IP are attenuated with aging. Much of this work has been performed in animal models or in human in vitro studies. Interestingly, no previous study directly examined the underlying mechanisms of this observation in humans using in vivo techniques. One potential explanation for an age-related reduction of the protective effect of IP relates to a direct effect on the endothelium.

Much scientific effort has been devoted to develop a human in vivo model to study ischemia and reperfusion injury. Recently, publications emerged using the flow mediated dilation (FMD) of the brachial or radial artery before and after a sustained ischaemic stimulus (20 minutes) to establish the presence of a blunted endothelial function after ischaemia reperfusion injury.3, 4 This effect of reperfusion injury on the endothelial function can be abrogated by ischemic preconditioning.3 Endothelial dysfunction is acknowledged to be the first (subclinical) manifestation of atherosclerosis and cardiovascular disease.5, 6 It is significantly correlated to occurrence of myocardial infarction and stroke.6 Assessment of the flow mediated dilation of the brachial artery as measure of endothelial (dys)function, is a validated model to research effects of possible protective strategies3, 4 and perform mechanistic experiments4, 7, 8 on IR-injury in humans in vivo.

Several previous studies failed to demonstrate the ability of pharmacological stimuli to mimic the beneficial effects of IP in aging vessels.9 Restoration of the age-related reduction in effectiveness of IP may be possible through exercise training. Indirect evidence indicates that physical activity, independent of other cardiovascular risk factors, protects against an occurrence as well as the severity of a myocardial infarction in humans.10 Although this suggests that physical activity may beneficially influence the age-related reduction in IP, no previous study provided direct evidence for this hypothesis in humans.

In this cross-sectional observational experiment we will study the impact of aging (young versus older subjects) and physical fitness (sedentary versus trained older subjects) on the protective effects of ischaemic preconditioning on brachial artery endothelial function after ischaemia-reperfusion injury in healthy humans in vivo.

We hypothesize that aging is associated with an attenuated ability of ischaemic preconditioning to prevent the decrease in brachial artery endothelial function observed after ischaemia reperfusion injury. Moreover, we expect that the age-related reduction in effectiveness of ischaemic preconditioning to prevent endothelial dysfunction after reperfusion injury is (at least partly) preserved in trained older subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young volunteers : age 18-30
* Healthy older volunteers: age >55 years
* Sedentary: <1 h exercise per week
* Trained: >5 h exercise per week
* All subjects: written informed consent

Exclusion Criteria:

* Smoking
* History of any cardiovascular disease
* Hypertension (in supine position: systole >140 mmHg, diastole >90 mmHg)
* Diabetes Mellitus (fasting glucose >7.0 mmol/L or random glucose >11.0 mmol/L)
* Hyperlipidaemia (fasting total cholesterol >6.5 mmol/L)
* Chronic use of medication known to interfere with the cardiovascular system
* Professional athletes
* BMI >30 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population: Young sedentary volunteers (n=23, age 18-30), young active volunteers (n=23, age 18-30), older sedentary subjects (n=23, >55 years) and older physically active subjects (n=23, >55 years).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
endothelial reperfusion injury | cross-sectional observation (single time point)
  Change in endothelial function (measured with flow mediated dilation) after ischaemia reperfusion injury (induced by 20 minutes ischemia) with and without precedence of ischaemic preconditioning (by 3 cycles of 5-minutes of ischaemia).

CONTACTS AND LOCATIONS:
Overall Officials: Dick Thijssen, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Department of Physiology, Nijmegen, Netherlands